CLINICAL TRIAL: NCT06258980
Title: Professor and Consultant of Pediatric Hematology Faculty of Medicine, Minia University, Al Minya, Egypt.
Brief Title: Use of Recombinant Factor VII as a Prophylactic Therapy for Adolescent Females With Heavy Menstrual Bleeding
Status: Completed | Type: Observational
Sponsor: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Gehan Lotfy Abdel Hakeem, professor of pediatric hematology, Minia University, Minia University Hospital
Other Study IDs: MiniaUH
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Assessing the Bleeding Profile and the Quality of Life of the Enrolled Patients Before and 1 Year After Drug Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- heavily menstruating females with glanzmannns Thrombaesthenia
  Interventions: Drug: Proph7

INTERVENTIONS:
Drug: Proph7 — Prophylactic recombinant FVII for heavily menorrhagic adolescent Glanzmanns Thrombaesthenia females

SUMMARY:
the study is conducted on adolescent females proved to be Glanzmanns Thrombaesthenia with heavy menstrual bleeding by the use of 3 doses of recombinant factor VII in the first day of their cycles. bleeding profile and quality of life were assessed before and 1year after this regular recombinant factor VII administration.

ELIGIBILITY:
Inclusion Criteria:

* adolescent females proved to be Glanzmanns Thrombaesthenia heavy menstrual bleeding no improvment by platelet transfusion or antifibrinolytic therapy

Exclusion Criteria:

chronic systemic disease previous allergic reaction to recombinant FVII

-

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — heavy menstrual bleeders
Study Population: adolescent females known Glanzmanns Thrombaesthenia with heavy menstrual bleeding
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
regular accepted menstrual cycles less than 6 days | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gehan Lotfy Abdel Hakeem, Al Minyā, Egypt

IPD SHARING:
Plan to Share IPD: No